CLINICAL TRIAL: NCT06073652
Title: Safety and Efficacy of a Starter Infant Formula With Synbiotics: a Double-blind, Randomized, Controlled Trial
Brief Title: Starter Infant Formula With Synbiotics
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Collaborators: Iqvia Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 21.14.INF
Record Dates: First submitted 2022-11-09; First posted 2023-10-10 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Healthy Infants

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: There are two masked, randomized formula-fed intervention groups, Control Formula (CF) and experimental Formula (EF)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control formula group (Active Comparator): The Control Formula group will receive 1st age infant formula exclusively for the first six months.
  Interventions: Other: Control 1st age starter infant formula
- Experimental formula group (Experimental): The Experimental Formula group will receive 1st age infant formula identical to Control formula, but supplemented with a HMO blend and a probiotic exclusively for the first six months.
  Interventions: Other: Experimental 1st age starter infant formula

INTERVENTIONS:
Other: Control 1st age starter infant formula — A standard bovine milk-based term infant formula.
  Arms: Control formula group
Other: Experimental 1st age starter infant formula — Same content as Control formula plus supplemented with a HMO blend and a probiotic
  Arms: Experimental formula group

SUMMARY:
This randomized, double-blind, controlled intervention trial aims to evaluate the safety and efficacy of a starter infant formula supplemented with an HMO blend and a probiotic, and will provide evidence on the safety and efficacy of the innovative prebiotic/ probiotic blend to support age-appropriate infant growth, a healthy gut microbiome, gastrointestinal (GI) tolerance and GI health, and immune development.

ELIGIBILITY:
Inclusion Criteria:

1. Evidence of personally signed and dated informed consent document indicating that at least one of the infant's parent(s)/LAR(s), as per local regulation, have been informed of all pertinent aspects of the study.
2. Infants whose parent(s)/LAR(s) have reached the legal age of majority in the countries where the study is conducted.
3. Able to temporarily store stool samples in a household freezer.
4. Infants whose parent(s)/LAR(s) are willing and able to comply with scheduled visits, and the requirements of the study protocol.
5. Infants whose parent(s)/LAR(s) are able to be contacted directly by telephone throughout the study.
6. Infants must meet all of the following inclusion criteria to be eligible for enrollment into the study:

   1. Healthy term infant (≥37 weeks of gestation).
   2. At enrollment visit, post-natal age ≥14 to ≤35 days / 0.75 - 1 month (date of birth = day 0)
   3. Birth weight ≥ 2500g and ≤ 4500g.
   4. For formula-fed groups, infants must be exclusively consuming and tolerating a cow's milk infant formula at time of enrollment and their parent(s)/LAR(s) must have independently elected, before enrollment, not to breastfeed.
   5. For the breastfed group, infants must have been exclusively consuming breastmilk since birth (small amounts of other feedings allowed during the first three days of life before breastfeeding is well-established), and their parent(s)/LAR(s) must have made the decision to continue exclusively breastfeeding until at least 4 months of age.

Exclusion Criteria:

1. Infants with conditions requiring infant feedings other than those specified in the protocol.
2. Infants who have a medical condition or history that could increase the risk associated with study participation or interfere with the interpretation of study results, including:

   1. Evidence of major congenital malformations (e.g., cleft palate, extremity malformation).
   2. Suspected or documented systemic or congenital infections (e.g., human immunodeficiency virus, cytomegalovirus, syphilis).
   3. Previous or ongoing severe medical or laboratory abnormality (acute or chronic) which, in the judgment of the investigator, would make the infant inappropriate for entry into the study. Of note, children who are normally healthy but at the time of enrolment suffering from acute illness in a minor condition which are common in childhood and do not require some of the exclusionary medication mentioned below can be enrolled.
3. Infants who are presently receiving or have received prior to enrolment any of the following: medication(s) or supplement(s) which are known or suspected to affect the following: fat digestion, absorption, and/or metabolism (e.g., pancreatic enzymes); stool microbiota and characteristics (e.g., oral, or systemic antibiotics, glycerin suppositories, bismuth-containing medications, docusate, Maltsupex, or lactulose); growth (e.g., insulin or growth hormone); gastric acid secretion.
4. Currently participating or having participated in another interventional clinical trial since birth.

Ages: 14 Days to 35 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 240 (Actual)
Dates: Start 2023-07-05 (Actual); Primary Completion 2024-08-14 (Actual); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Safety of experimental formula demonstrated by growth | Baseline Visit 1 to 4 months of age Visit 5
  Weight gain comparison between infants from experimental and control group

SECONDARY OUTCOMES:
Efficacy of experimental formula demonstrated by fecal sIgA concentration. | Baseline Visit 1 to 4 months of age Visit 5
  Concentration of sIgA in fecal samples
Fecal microbiome | Baseline Visit 1 to 6 month of age Visit 6
  Fecal microbiota modulating effect
Fecal metabolic profile | Baseline Visit 1 to 6 month of age Visit 6
  Fecal pH, fecal organic acids measurement from fecal samples
Fecal markers of immune health and gut barrier function | Baseline Visit 1 to 6 month of age Visit 6
  Fecal markers of immune health and gut barrier, such as but not restricted to calprotectin and α-1-antitrypsin assessed by ELISA.
Fecal cytokine profile | Baseline Visit 1 to 6 month of age Visit 6
  Fecal cytokine profile (such as but not restricted to: IL-6, IL-8, IL-1b, IL-22, IFN-γ) using multiplex assays.
Blood markers of systemic immunity | Baseline Visit 1 to 4 months of age Visit 5
  Immunotyping and plasma immune proteomics and Vaccine specific antibodies measurement from blood samples
3-day GI Symptom and Behavior Diary | Baseline Visit 1 to 6 month of age Visit 6
  GI tolerance, GI symptoms and GI-related behaviors
Infant Gastrointestinal Symptom Questionnaire (IGSQ-13) Index questionnaire | Baseline Visit 1 to 6 month of age Visit 6
  GI tolerance, GI symptoms and GI-related behaviors
Weight (g) | Baseline Visit 1 to 6 month of age Visit 6
  Anthropometric measurement. Weight and height will be combined to report BMI in kg/m^2
Length (cm) | Baseline Visit 1 to 6 month of age Visit 6
  Anthropometric measurement. Weight and height will be combined to report BMI in kg/m^2
Head circumference (cm) | Baseline Visit 1 to 6 month of age Visit 6
  Anthropometric measurement
Respiration | Baseline Visit 1 to 6 month of age Visit 6
  Vital signs
Heart rate | Baseline Visit 1 to 6 month of age Visit 6
  Vital signs
Body temperature | Baseline Visit 1 to 6 month of age Visit 6
  Vital signs
Physical examination | Baseline Visit 1 to 3 years of age Observational Follow Up Visit 5
  Infant illness and infection outcomes
Pediatric Immune System Index and Infant Illness Questionnaire | Baseline Visit 1 to 3 years of age Observational Follow Up Visit 5
  Infant illness and infection outcomes
Antibiotic and antipyretic use | Baseline Visit 1 to 6 month of age Phone visit 7
  Concomitant medication reporting

CONTACTS AND LOCATIONS:
Overall Officials: Maria Rosario Capeding, Dr, Principal Investigator — Asian Hospital Medical Center; Mitzi Trinidad Aseron, Dr, Principal Investigator — University of Perpetual Help Dalta Medical Center; Vinna Marie Quinones, Dr, Principal Investigator — University of the East Ramon Magsaysay Memorial Medical Center
Locations (3):
- Philippines (3):
  - Asian Hospital and Medical Center, Manila
  - University of Perpetual Help DALTA Medical Center, Manila
  - University of the East Ramon Magsaysay Memorial Medical Center, Manila